CLINICAL TRIAL: NCT01170663
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase 3 Study of Weekly Paclitaxel With or Without Ramucirumab (IMC-1121B) Drug Product in Patients With Metastatic Gastric Adenocarcinoma, Refractory to or Progressive After First-Line Therapy With Platinum and Fluoropyrimidine
Brief Title: A Study of Paclitaxel With or Without Ramucirumab (IMC-1211B) in Metastatic Gastric Adenocarcinoma
Acronym: RAINBOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13894; I4T-IE-JVBE (Other: Eli Lilly and Company); CP12-0922 (Other: ImClone Systems); 2010-020426-18 (EudraCT Number)
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
Keywords: Metastatic Adenocarcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramucirumab (IMC-1211B) Drug Product (DP) and Paclitaxel (Experimental): Ramucirumab (IMC-1211B) DP and Paclitaxel
  Interventions: Biological: Ramucirumab (IMC-1211B) DP; Drug: Paclitaxel
- Placebo and Paclitaxel (Placebo Comparator): Placebo and Paclitaxel
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Biological: Ramucirumab (IMC-1211B) DP — 8 milligrams/kilogram (mg/kg) intravenous (IV) infusion on Days 1 and 15 of every 4-week cycle
  Other Names: LY3009806; IMC-1211B
  Arms: Ramucirumab (IMC-1211B) Drug Product (DP) and Paclitaxel
Drug: Placebo — Ramucirumab placebo IV infusion on Days 1 and 15 of every 4-week cycle
  Arms: Placebo and Paclitaxel
Drug: Paclitaxel — Paclitaxel 80 milligrams per square meter (mg/m²) IV infusion on Days 1, 8, and 15 of every 4-week cycle

SUMMARY:
This is a Phase III randomized multicenter double-blind, placebo controlled trial evaluating the safety and efficacy of paclitaxel plus ramucirumab (IMC-1211B) drug product (DP) compared to paclitaxel plus placebo.

DETAILED DESCRIPTION:
The aim of this study is to determine if paclitaxel given together with ramucirumab (IMC-1211B) as second line therapy will prolong overall survival (OS) compared to paclitaxel alone.

Approximately 663 participants (at least 18 years) in approximately 200 study centers and in approximately 30 countries will be randomized with histologically or cytologically confirmed metastatic gastric or gastroesophageal junction adenocarcinoma. Participants must have received at least one cycle of first line therapy with any platinum/fluoropyrimidine doublet with or without anthracycline (epirubicin or doxorubicin) and must have discontinued this therapy prior to study entry due to disease progression.

Upon registration and completion of screening procedure and reviewing the Inclusion and Exclusion Criteria eligible participants will be randomized to receive either paclitaxel plus ramucirumab or paclitaxel plus placebo.

Ramucirumab (IMC-1211B) DP/placebo will be administered IV on Days 1 and 15, paclitaxel will be administered IV on Days 1, 8 and 15 of a 4 weekly cycle.

Participants will be continuously treated and monitored until radiographic or symptomatic progression of disease, toxicity requiring cessation, protocol noncompliance, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma
* Metastatic disease or locally advanced, unresectable disease
* Disease progression during or within 4 months after the last dose of the first-line therapy (platinum/fluoropyrimidine doublet with or without anthracycline)
* Organs are functioning well (liver, kidney, blood)
* Good performance status Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1

Exclusion Criteria:

* First line chemotherapy for metastatic gastric cancer other than platinum/fluoropyrimidine doublet with or without anthracycline
* Previous systemic therapy with other anti-angiogenic drugs
* Uncontrolled high blood pressure
* Symptomatic or poorly controlled heart disease or had a heart attack or stroke within the last 6 month
* Evidence of central nervous system (CNS) metastasis at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2010-12; Primary Completion 2013-07 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (159):
- United States (13):
  - ImClone Investigational Site, Burbank, California
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Miramar, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Honolulu, Hawaii
  - ImClone Investigational Site, East Orange, New Jersey
  - ImClone Investigational Site, Albuquerque, New Mexico
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Chattanooga, Tennessee
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Seattle, Washington
- Argentina (4):
  - ImClone Investigational Site, Buenos Aires
  - ImClone Investigational Site, Caba
  - ImClone Investigational Site, Rosario
  - ImClone Investigational Site, Santa Fe
- Australia (10):
  - ImClone Investigational Site, Bankstown, New South Wales
  - ImClone Investigational Site, Kogarah, New South Wales
  - ImClone Investigational Site, Liverpool, New South Wales
  - ImClone Investigational Site, Wollongong, New South Wales
  - ImClone Investigational Site, Southport, Queensland
  - ImClone Investigational Site, Kurralta Park, South Australia
  - ImClone Investigational Site, Coburg, Victoria
  - ImClone Investigational Site, Footscray, Victoria
  - ImClone Investigational Site, Frankston, Victoria
  - ImClone Investigational Site, Parkville, Victoria
- Austria (4):
  - ImClone Investigational Site, Graz
  - ImClone Investigational Site, Linz
  - ImClone Investigational Site, Steyr
  - ImClone Investigational Site, Vienna
- Belgium (5):
  - ImClone Investigational Site, Bonheiden
  - ImClone Investigational Site, Bruges
  - ImClone Investigational Site, Brussels
  - ImClone Investigational Site, Edegem
  - ImClone Investigational Site, Leuven
- Brazil (16):
  - ImClone Investigational Site, Belo Horizonte
  - ImClone Investigational Site, Caxias do Sul
  - ImClone Investigational Site, Dois Lajeados
  - ImClone Investigational Site, Gávea
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Itajaí
  - ImClone Investigational Site, Londrina
  - ImClone Investigational Site, Passo Fundo
  - ImClone Investigational Site, Porto Alegre
  - ImClone Investigational Site, Porto Alegre-Rs
  - ImClone Investigational Site, Ribeirão Preto
  - ImClone Investigational Site, Rio de Janeiro
  - ImClone Investigational Site, Salvador
  - ImClone Investigational Site, Sao Jose Rio Preto
  - ImClone Investigational Site, São Paulo
  - ImClone Investigational Site, Sorocaba
- Bulgaria (2):
  - ImClone Investigational Site, Sofia
  - ImClone Investigational Site, Varna
- Chile (2):
  - ImClone Investigational Site, Providencia
  - ImClone Investigational Site, Viña del Mar
- ImClone Investigational Site, Tallinn, Estonia
- France (8):
  - ImClone Investigational Site, Besançon
  - ImClone Investigational Site, Brest
  - ImClone Investigational Site, Clermont-Ferrand
  - ImClone Investigational Site, Marseille
  - ImClone Investigational Site, Montbéliard
  - ImClone Investigational Site, Montpellier
  - ImClone Investigational Site, Paris
  - ImClone Investigational Site, Saint-Etienne
- Germany (12):
  - ImClone Investigational Site, Berlin
  - ImClone Investigational Site, Bielefeld
  - ImClone Investigational Site, Dresden
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Frankfurt
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Heidelberg
  - ImClone Investigational Site, Leipzig
  - ImClone Investigational Site, Mainz
  - ImClone Investigational Site, Munich
  - ImClone Investigational Site, Recklinghausen
  - ImClone Investigational Site, Tübingen
- Hungary (5):
  - ImClone Investigational Site, Budapest
  - ImClone Investigational Site, Gyula
  - ImClone Investigational Site, Kaposvár
  - ImClone Investigational Site, Pécs
  - ImClone Investigational Site, Székesfehérvár
- Israel (7):
  - ImClone Investigational Site, Beersheba
  - ImClone Investigational Site, Haifa
  - ImClone Investigational Site, Holon
  - ImClone Investigational Site, Jerusalem
  - ImClone Investigational Site, Petah Tikva
  - ImClone Investigational Site, Tel Aviv
  - ImClone Investigational Site, Tel Litwinsky
- Italy (9):
  - ImClone Investigational Site, Ancona
  - ImClone Investigational Site, Bari
  - ImClone Investigational Site, Bergamo
  - ImClone Investigational Site, Catania
  - ImClone Investigational Site, Genova
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Padua
  - ImClone Investigational Site, Pisa
  - ImClone Investigational Site, Torino
- Japan (13):
  - ImClone Investigational Site, Aichi
  - ImClone Investigational Site, Chiba
  - ImClone Investigational Site, Ehime
  - ImClone Investigational Site, Fukuoka
  - ImClone Investigational Site, Hokkaido
  - ImClone Investigational Site, Kochi
  - ImClone Investigational Site, Osaka
  - ImClone Investigational Site, Osaka-Pref
  - ImClone Investigational Site, Ōita
  - ImClone Investigational Site, Saitama
  - ImClone Investigational Site, Shizuoka
  - ImClone Investigational Site, Tochigi
  - ImClone Investigational Site, Tokyo
- Lithuania (2):
  - ImClone Investigational Site, Kaunas
  - ImClone Investigational Site, Klaipėda
- Mexico (2):
  - ImClone Investigational Site, Juchitán
  - ImClone Investigational Site, Nuevo León
- Poland (7):
  - ImClone Investigational Site, Brzozów
  - ImClone Investigational Site, Bydgoszcz
  - ImClone Investigational Site, Gdansk
  - ImClone Investigational Site, Lodz
  - ImClone Investigational Site, Lublin
  - ImClone Investigational Site, Poznan
  - ImClone Investigational Site, Warsaw
- Portugal (5):
  - ImClone Investigational Site, Aveiro
  - ImClone Investigational Site, Coimbra
  - ImClone Investigational Site, Evora
  - ImClone Investigational Site, Porto
  - ImClone Investigational Site, Santa Maria da Feira
- Romania (4):
  - ImClone Investigational Site, Baia Mare
  - ImClone Investigational Site, Bucharest
  - ImClone Investigational Site, Iași
  - ImClone Investigational Site, Târgu Mureş
- Russia (5):
  - ImClone Investigational Site, Krasnodar
  - ImClone Investigational Site, Moscow
  - ImClone Investigational Site, Perm
  - ImClone Investigational Site, Saint Petersburg
  - ImClone Investigational Site, Ufa
- ImClone Investigational Site, Singapore, Singapore
- South Korea (4):
  - ImClone Investigational Site, Incheon
  - ImClone Investigational Site, Seongnam-si
  - ImClone Investigational Site, Seoul
  - ImClone Investigational Site, Suwon
- Spain (8):
  - ImClone Investigational Site, Ávila
  - ImClone Investigational Site, Burgos
  - ImClone Investigational Site, Jerez de la Frontera
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Majadahonda
  - ImClone Investigational Site, Palma de Mallorca
  - ImClone Investigational Site, Sabadell
  - ImClone Investigational Site, Seville
- Taiwan (6):
  - ImClone Investigational Site, Changhua
  - ImClone Investigational Site, Kaohsiung City
  - ImClone Investigational Site, Liouying/Tainan
  - ImClone Investigational Site, Taichung
  - ImClone Investigational Site, Tainan
  - ImClone Investigational Site, Taipei
- United Kingdom (4):
  - ImClone Investigational Site, Maidstone, Kent
  - ImClone Investigational Site, Guildford, Surrey
  - ImClone Investigational Site, Sutton, Surrey
  - ImClone Investigational Site, Wolverhampton, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ogata T, Narita Y, Wainberg ZA, Van Cutsem E, Yamaguchi K, Piao Y, Zhao Y, Peterson PM, Wijayawardana SR, Abada P, Chatterjee A, Muro K. Exploratory Analysis of Patients With Gastric/Gastroesophageal Junction Adenocarcinoma With or Without Liver Metastasis From the Phase 3 RAINBOW Study. J Gastric Cancer. 2023 Apr;23(2):289-302. doi: 10.5230/jgc.2023.23.e15. PMID 37129153
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Yamaguchi K, Shimada Y, Hironaka S, Sugimoto N, Komatsu Y, Nishina T, Omuro Y, Tamura T, Piao Y, Homma G, Jen MH, Liepa AM, Muro K. Quality of Life Associated with Ramucirumab Treatment in Patients with Advanced Gastric Cancer in Japan: Exploratory Analysis from the Phase III RAINBOW Trial. Clin Drug Investig. 2021 Jan;41(1):53-64. doi: 10.1007/s40261-020-00979-3. Epub 2020 Dec 23. PMID 33355909
- [Derived] Cascinu S, Bodoky G, Muro K, Van Cutsem E, Oh SC, Folprecht G, Ananda S, Girotto G, Wainberg ZA, Miron MLL, Ajani J, Wei R, Liepa AM, Carlesi R, Emig M, Ohtsu A. Tumor Response and Symptom Palliation from RAINBOW, a Phase III Trial of Ramucirumab Plus Paclitaxel in Previously Treated Advanced Gastric Cancer. Oncologist. 2021 Mar;26(3):e414-e424. doi: 10.1002/onco.13623. Epub 2020 Dec 23. PMID 33274542
- [Derived] De Vita F, Borg C, Farina G, Geva R, Carton I, Cuku H, Wei R, Muro K. Ramucirumab and paclitaxel in patients with gastric cancer and prior trastuzumab: subgroup analysis from RAINBOW study. Future Oncol. 2019 Aug;15(23):2723-2731. doi: 10.2217/fon-2019-0243. Epub 2019 Jun 25. PMID 31234645
- [Derived] Chau I, Fuchs CS, Ohtsu A, Barzi A, Liepa AM, Cui ZL, Hsu Y, Al-Batran SE. Association of quality of life with disease characteristics and treatment outcomes in patients with advanced gastric cancer: Exploratory analysis of RAINBOW and REGARD phase III trials. Eur J Cancer. 2019 Jan;107:115-123. doi: 10.1016/j.ejca.2018.11.013. Epub 2018 Dec 14. PMID 30557792
- [Derived] Tabernero J, Ohtsu A, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Ajani JA, Tomasek J, Safran H, Chandrawansa K, Hsu Y, Heathman M, Khan A, Ni L, Melemed AS, Gao L, Ferry D, Fuchs CS. Exposure-Response Analyses of Ramucirumab from Two Randomized, Phase III Trials of Second-line Treatment for Advanced Gastric or Gastroesophageal Junction Cancer. Mol Cancer Ther. 2017 Oct;16(10):2215-2222. doi: 10.1158/1535-7163.MCT-16-0895. Epub 2017 Jul 17. PMID 28716815
- [Derived] Al-Batran SE, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov ON, Kim TY, Cunningham D, Rougier P, Muro K, Liepa AM, Chandrawansa K, Emig M, Ohtsu A, Wilke H. Quality-of-life and performance status results from the phase III RAINBOW study of ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated gastric or gastroesophageal junction adenocarcinoma. Ann Oncol. 2016 Apr;27(4):673-9. doi: 10.1093/annonc/mdv625. Epub 2016 Jan 7. PMID 26747859
- [Derived] Shitara K, Muro K, Shimada Y, Hironaka S, Sugimoto N, Komatsu Y, Nishina T, Yamaguchi K, Segawa Y, Omuro Y, Tamura T, Doi T, Yukisawa S, Yasui H, Nagashima F, Gotoh M, Esaki T, Emig M, Chandrawansa K, Liepa AM, Wilke H, Ichimiya Y, Ohtsu A. Subgroup analyses of the safety and efficacy of ramucirumab in Japanese and Western patients in RAINBOW: a randomized clinical trial in second-line treatment of gastric cancer. Gastric Cancer. 2016 Jul;19(3):927-38. doi: 10.1007/s10120-015-0559-z. Epub 2015 Oct 28. PMID 26510663
- [Derived] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants that discontinued study drugs either due to progressive disease (PD), due to an adverse event or died due to any cause, but not necessarily had any survival-FU assessment done.
Groups:
- Ramucirumab (IMC-1211B) Plus Paclitaxel: 8 milligrams/kilogram (mg/kg) of ramucirumab (IMC-1121B) was administered by intravenous (IV) infusion on Days 1 and 15 in combination with 80 milligrams/square meter (mg/m²) paclitaxel administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle.
- Placebo Plus Paclitaxel: Placebo was administered by IV infusion on Days 1 and 15, in combination with 80 mg/m² paclitaxel administered on Days 1, 8, and 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Started (One participant randomized to placebo/paclitaxel arm but received ramucirumab (IMC-1121B) in error.) | 330 (Participant was included in ramucirumab (IMC-1121B)/paclitaxel treatment arm (safety population).) | 335 (Participant was included in the placebo/paclitaxel treatment arm (intent-to-treat (ITT) population).)
Received Any Treatment (Safety Pop) | 327 | 329
Completed | 316 | 315
Not Completed | 14 | 20
Not completed — Lost to Follow-up | 3 | 9
Not completed — Withdrawal of consent without follow-up | 11 | 11

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab (IMC-1211B) Plus Paclitaxel: 8 mg/kg of ramucirumab (IMC-1121B) was administered by IV infusion on Days 1 and 15 in combination with 80 mg/m² paclitaxel administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel | Total
Number analyzed (Participants) | 330 | 335 | 665
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 205 | 213 | 418
  >=65 years | 125 | 122 | 247
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 83] | 61 [24 to 84] | 61 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 92 | 193
  Male | 229 | 243 | 472
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 26 | 57
  Not Hispanic or Latino | 299 | 309 | 608
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 110 | 121 | 231
  Black or African American | 6 | 6 | 12
  White | 208 | 199 | 407
  More than one race | 0 | 1 | 1
  Other | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 2 | 0 | 2
  United States | 12 | 12 | 24
  Estonia | 5 | 5 | 10
  Taiwan | 14 | 16 | 30
  Spain | 8 | 13 | 21
  Russia | 8 | 13 | 21
  Chile | 1 | 3 | 4
  Italy | 13 | 15 | 28
  France | 20 | 14 | 34
  Australia | 18 | 23 | 41
  South Korea | 23 | 22 | 45
  Lithuania | 6 | 6 | 12
  Austria | 4 | 2 | 6
  United Kingdom | 6 | 9 | 15
  Hungary | 20 | 9 | 29
  Mexico | 2 | 2 | 4
  Argentina | 1 | 0 | 1
  Poland | 15 | 18 | 33
  Brazil | 19 | 16 | 35
  Belgium | 12 | 14 | 26
  Singapore | 2 | 3 | 5
  Romania | 7 | 7 | 14
  Bulgaria | 7 | 5 | 12
  Germany | 20 | 20 | 40
  Japan | 68 | 72 | 140
  Hong Kong | 2 | 1 | 3
  Israel | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time (OS)
Description: OS time was measured from date of randomization to date of death from any cause. Participants who were not known to have died on or before the date of data cut-off, OS data was censored on the last date (on or before the cut-off date) the participant was known to be alive.
Time Frame: Randomization up to 27.5 months
Population: All participants according to the treatment group to which they were randomized. Participants censored: Ramucirumab (IMC-1211B) plus Paclitaxel =74, Placebo plus Paclitaxel =75.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 330 | 335
months | 9.6 [8.5 to 10.8] | 7.4 [6.3 to 8.4]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1211B) Plus Paclitaxel vs Placebo Plus Paclitaxel; Test type: Superiority or Other; p = 0.0169, Stratified Log Rank Test; Adjusted for stratification factors: geographic region, time-to-progression from start of first-line therapy and disease measurability; Hazard Ratio (HR) = 0.807, 95% CI 2-sided [0.678 to 0.962]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was measured from date of randomization to first radiographically documented progressive disease (PD) or death due to any cause. PD defined using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm. Participants who had no baseline or post baseline radiological tumor assessment were censored at date of randomization. Participants who had no tumor progression or death within 2 scan intervals following the last assessment were censored at the date of last radiographic tumor assessment. Participants who began new anticancer treatment and had no tumor progression were censored at date of assessment prior to initiation of new therapy. Participants lost to follow-up or withdrew consent were censored at the date of their last assessment.
Time Frame: Randomization up to 22.2 months
Population: All participants according to the treatment group to which they were randomized. Participants censored: Ramucirumab (IMC-1211B) plus Paclitaxel =51, Placebo plus Paclitaxel =39.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 330 | 335
months | 4.4 [4.2 to 5.3] | 2.9 [2.8 to 3.0]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1211B) Plus Paclitaxel vs Placebo Plus Paclitaxel; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.635, 95% CI 2-sided [0.536 to 0.752]

3. Secondary Outcome: Time to Progressive Disease (TTP)
Description: TTP was defined as the time from randomization until date of radiographic progression using RECIST v1.1 criteria. PD was defined as having a ≥20% increase in sum of longest diameter (LD) of target lesions and at minimum 5 millimeters (mm) increase above nadir. Participants who did not progress or were lost to follow-up were censored at the date of last tumor assessment. Participants who had no baseline tumor assessment or no post baseline assessment and no death reported with 2 scan intervals post randomization were censored at date of randomization. Participants with no progression and not died within 2 scan intervals after last assessment were censored at date of last tumor assessment. Participants with no post baseline assessment or tumor progression but death reported within 2 scan intervals after randomization were censored at date of death.
Time Frame: Baseline up to 22.2 months
Population: All participants according to the treatment group to which they were randomized. Participants censored: Ramucirumab (IMC-1211B) plus Paclitaxel =107, Placebo plus Paclitaxel =94.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 330 | 335
months | 5.52 [4.50 to 5.68] | 3.02 [2.86 to 4.14]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1211B) Plus Paclitaxel vs Placebo Plus Paclitaxel; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.596, 95% CI 2-sided [0.494 to 0.720]

4. Secondary Outcome: Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or PD
Description: BOR was defined as the best response across all time points from randomization until radiologically confirmed PD using RECIST, v1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions. PR was defined as having a ≥30% decrease in sum of LD of target lesions. PD was defined as having a ≥20% increase in sum of LD of target lesions and ≥5 mm increase above nadir. SD was defined as small changes that did not meet above criteria.
Time Frame: Randomization up to 22.2 months
Population: All participants according to the treatment group to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 330 | 335
percentage of participants
  CR | 0.6 | 0.3
  PR | 27.3 | 15.8
  SD | 52.1 | 47.5
  PD | 13.0 | 24.8
  Not Evaluable | 0.3 | 0.9
  No Tumor Response Evaluation | 6.7 | 10.7

5. Secondary Outcome: Percentage of Participants With CR or PR (Objective Response Rate [ORR])
Description: ORR was the percentage of participants who had CR or PR defined using RECIST v1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions. PR was defined as having a ≥30% decrease in sum of LD of target lesions. Percentage of participants calculated as: (number of participants with CR + PR)/(total number of participants)*100.
Time Frame: Randomization up to 22.2 months
Population: All participants according to the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 330 | 335
percentage of participants | 27.9 [23.3 to 33.0] | 16.1 [12.6 to 20.4]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1211B) Plus Paclitaxel vs Placebo Plus Paclitaxel; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Adjusted for stratification factors: geographic region, time-to-progression from the start of first-line therapy and disease measurability; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.45 to 3.16]

6. Secondary Outcome: Percentage of Participants With Anti-Ramucirumab Antibodies (Serum Anti-Ramucirumab Antibody Assessment )(Immunogenicity)
Description: Participants who developed treatment-emergent antibody responses to Ramucirumab (IMC-1121B) after baseline.
Time Frame: Prior to and after ramucirumab (IMC-1121B) infusion: Day 1 Cycles 1, 2 and 3 (28-day cycles) Doses 1, 4, 7 and 30-37 days after last dose of study therapy up to 103 weeks
Population: All participants according to the treatment group to which they were randomized and received at least 1 dose of study drug with anti-ramucirumab antibodies.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 320 | 323
percentage of participants | 1.6 | 0.3

7. Secondary Outcome: Maximum Concentration (Cmax) After First Ramucirumab (IMC-1211B) Infusion
Time Frame: Cycle 1, Day 1, 1 hour post end of infusion (28-day cycles)
Population: All participants who received Ramucirumab (IMC-1121B) plus Paclitaxel and had Cmax observations at specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 259
micrograms/milliliter (µg/mL) | 146 (28)

8. Secondary Outcome: Cmax After 4th Ramucirumab (IMC-1211B) Infusion
Time Frame: Cycle 2, Day 15 1 hour post end of infusion (28-day cycles)
Population: All participants who received Ramucirumab (IMC-1121B) plus Paclitaxel and had Cmax observations at specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 200
µg/mL | 193 (34)

9. Secondary Outcome: Cmax After 7th Ramucirumab (IMC-1211B) Infusion
Time Frame: Cycle 4, Day 1, 1 hour post end of infusion (28-day cycles)
Population: All participants who received Ramucirumab (IMC-1121B) plus Paclitaxel and had Cmax observations at specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 127
µg/mL | 216 (30)

10. Secondary Outcome: Minimum Concentration (Cmin) Prior to First Ramucirumab (IMC-1211B) Infusion
Description: This outcome measure was included in error as the time point was before ramucirumab (IMC-1211B) was administered. Cmin was not analyzed.
Time Frame: Cycle 1, Day 1 predose (28-day cycles)
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 0

11. Secondary Outcome: Cmin Prior to 4th Ramucirumab (IMC-1211B) Infusion
Time Frame: Cycle 2, Day 15 (28-day cycle)
Population: All participants who received Ramucirumab (IMC-1121B) plus Paclitaxel and had Cmin observations at specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 203
µg/mL | 45.0 (50)

12. Secondary Outcome: Cmin Prior to 7th Ramucirumab (IMC-1211B) Infusion
Time Frame: Cycle 4, Day 1 (28-day cycles)
Population: All participants who received Ramucirumab (IMC-1121B) plus Paclitaxel and had Cmin observations at specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel
Number analyzed (Participants) | 142
µg/mL | 62.8 (47)

13. Secondary Outcome: Change From Baseline to End of Therapy in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life: Questionnaire (QLQ-C30) in Global Health Status
Description: EORTC QLQ-C30 v3.0 is a 30-item, self-administered questionnaire with multidimensional scales assessing 15 domains (5 functional domains [physical, role, cognitive, emotional, and social], 9 symptom scales [fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties] and global health status scale). 28 questions assessed on a 1 (not at all) to 4 (very much) scale and the remaining 2 questions used a 1 (poor) to 7 (excellent) scale. A linear transformation was applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For the functional domains and global health status scale, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms.
Time Frame: Baseline, end of therapy (up to 103 weeks)
Population: All participants according to the treatment group to which they were randomized with baseline and end of treatment Global Health Status observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 209 | 202
units on a scale | -13.5 (23.24) | -12.1 (24.81)
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1211B) Plus Paclitaxel vs Placebo Plus Paclitaxel; Test type: Superiority or Other; p = 0.3973, ANCOVA — Analysis of covariance (ANCOVA) included treatment group, randomization stratification factors and baseline value of Global Health Status scale

14. Secondary Outcome: Change From Baseline to End of Therapy in European Quality of Life Questionnaire-5 Dimension (EuroQol EQ-5D) Index Score
Description: The EQ-5D is a generic, multidimensional, health status instrument. The profile allowed participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale [1 (no problem), 2 (some problems), and 3 (major problems)]. These combinations of responses were converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension). A negative change indicated a worsening of the participant's health status.
Time Frame: Baseline, end of therapy (up to 103 weeks)
Population: All participants according to the treatment group to which they were randomized with baseline and end of treatment EQ-5D observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 205 | 201
units on a scale | -0.16 (0.279) | -0.19 (0.337)

15. Other Pre Specified Outcome: Number of Participants With Serious and Other Non-serious Adverse Events (AE) and Who Died
Description: Participants who died or who had clinically significant events defined as serious AEs (SAEs) and other non-serious AEs (regardless of causality). A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to 103 weeks and within 30 days of last dose of study drug
Population: All randomized participants who received at least 1 dose of study drug and based on the treatment each participant received.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1211B) Plus Paclitaxel | Placebo Plus Paclitaxel
Number analyzed (Participants) | 327 | 329
participants
  SAEs | 161 | 146
  Other Non-serious AEs | 324 | 321
  Died | 37 | 52

ADVERSE EVENTS:
Description: One (1) participant was randomized to the placebo group but received ramucirumab in error. This participant was included in the ramucirumab group in the Safety population (as treated).
Groups:
- Ramucirumab and Paclitaxel: 8 mg/kg ramucirumab (IMC1121B) was administered by IV infusion on Days 1 and 15 in combination with 80 mg/m² administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle.
- Placebo and Paclitaxel: Placebo was administered by IV infusion on Days 1 and 15, in combination with 80 mg/m² administered on Days 1, 8, and 15 of a 28-day cycle.
Arm/Group | Ramucirumab and Paclitaxel | Placebo and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 161/327 | 146/329
Other Adverse Events (participants affected / at risk) | 324/327 | 321/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab and Paclitaxel (N=327) | Placebo and Paclitaxel (N=329)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 7 (10)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 12 (17) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 11 (12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 5 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 3 (3)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (3) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 5 (6)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 4 (5)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 10 (11)
Asthenia (General disorders) | 5 (7) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 2 (2)
Drowning (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 7 (9)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 8 (10) | 9 (12)
Injection site injury (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 7 (9)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3)
Device related infection (Infections and infestations) | 2 (2) | 3 (3)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 3 (6) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (7) | 4 (5)
Septic shock (Infections and infestations) | 3 (3) | 1 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 6 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 (65) | 49 (66)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (2)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1/226 (1) | 0/237 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Paclitaxel (N=327) | Placebo and Paclitaxel (N=329)
Anaemia (Blood and lymphatic system disorders) | 110 (261) | 116 (274)
Leukopenia (Blood and lymphatic system disorders) | 111 (471) | 69 (199)
Neutropenia (Blood and lymphatic system disorders) | 174 (878) | 102 (247)
Thrombocytopenia (Blood and lymphatic system disorders) | 43 (103) | 20 (37)
Abdominal distension (Gastrointestinal disorders) | 20 (27) | 20 (25)
Abdominal pain (Gastrointestinal disorders) | 98 (165) | 62 (104)
Abdominal pain upper (Gastrointestinal disorders) | 31 (48) | 35 (52)
Ascites (Gastrointestinal disorders) | 31 (46) | 25 (39)
Constipation (Gastrointestinal disorders) | 70 (95) | 71 (89)
Diarrhoea (Gastrointestinal disorders) | 105 (250) | 76 (126)
Dysphagia (Gastrointestinal disorders) | 17 (25) | 17 (18)
Nausea (Gastrointestinal disorders) | 114 (236) | 106 (183)
Stomatitis (Gastrointestinal disorders) | 64 (103) | 24 (33)
Vomiting (Gastrointestinal disorders) | 85 (142) | 65 (111)
Asthenia (General disorders) | 68 (179) | 45 (73)
Fatigue (General disorders) | 128 (281) | 104 (209)
Oedema peripheral (General disorders) | 82 (122) | 45 (57)
Pyrexia (General disorders) | 56 (83) | 35 (53)
Nasopharyngitis (Infections and infestations) | 23 (34) | 19 (24)
Urinary tract infection (Infections and infestations) | 18 (22) | 11 (11)
Alanine aminotransferase increased (Investigations) | 20 (43) | 18 (22)
Aspartate aminotransferase increased (Investigations) | 27 (62) | 17 (23)
Weight decreased (Investigations) | 45 (79) | 49 (68)
Decreased appetite (Metabolism and nutrition disorders) | 131 (225) | 105 (172)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 31 (47) | 13 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (23) | 9 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (54) | 20 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 38 (48) | 39 (47)
Myalgia (Musculoskeletal and connective tissue disorders) | 34 (62) | 32 (44)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (21) | 10 (10)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 26 (26)
Dizziness (Nervous system disorders) | 20 (25) | 13 (16)
Dysgeusia (Nervous system disorders) | 29 (32) | 21 (23)
Headache (Nervous system disorders) | 32 (50) | 22 (37)
Neuropathy peripheral (Nervous system disorders) | 47 (88) | 30 (51)
Paraesthesia (Nervous system disorders) | 24 (41) | 25 (41)
Peripheral sensory neuropathy (Nervous system disorders) | 57 (122) | 36 (63)
Polyneuropathy (Nervous system disorders) | 18 (31) | 22 (38)
Insomnia (Psychiatric disorders) | 31 (32) | 26 (27)
Proteinuria (Renal and urinary disorders) | 55 (156) | 20 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (46) | 26 (35)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 9 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (61) | 31 (38)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 100 (157) | 23 (34)
Alopecia (Skin and subcutaneous tissue disorders) | 107 (137) | 127 (159)
Dry skin (Skin and subcutaneous tissue disorders) | 25 (28) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (23) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 35 (44) | 25 (28)
Hypertension (Vascular disorders) | 78 (155) | 16 (25)

LIMITATIONS AND CAVEATS:
One (1) participant was randomized to the placebo/paclitaxel group but received ramucirumab in error. For ITT population this participant was included in placebo/paclitaxel group and for the Safety population included in the ramucirumab group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.